CLINICAL TRIAL: NCT02061033
Title: GLOBAL HEMOSTATIC METHODS IN HEMOPHILIA AND VON WILLEBRAND'S DISEASE CORRELATION WITH PATIENTS' CLINICAL STATUS AND USEFULNESS FOR TREATMENT MONITORING
Brief Title: Global Hemostatic Methods in Hemophilia and Von Willebrand's Disease
Acronym: GHMHW
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: The Swedish Society of Medicine (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jovan P. Antovic MD, PhD, Associate professor, Consultant, Karolinska University Hospital
Other Study IDs: GHMJA2014
Record Dates: First submitted 2014-02-07; First posted 2014-02-12 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Hemophilia A; Hemophilia B; Von Willebrand's Disease
Keywords: Hemophilia A; Hemophilia B; Von Willebrand's Disease; Endogen thrombin potential; Overall hemostatic potential; Microparticles; Fibrin clot
MeSH Terms: conditions — Hemophilia A; Hemophilia B; von Willebrand Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Citrated plasma and whole blood DNA samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with hemophilia who have the same level of deficient factor(s) may express different severity of clinical presentation and bleeding tendency. Therefore a test which could determine overall hemostasis rather than simple concentration of a single deficient factor may correlate better with clinical phenotype in these patients.

The investigators will therefore study the usefulness of global hemostatic methods (endogenous thrombin potential (ETP), overall hemostatic potential (OHP), fibrin clot structure) and microparticles in the prediction of severity of bleeding and estimation of response to the treatment in patients with hemophilia.

Since hemophilia patients on prophylactic treatment virtually do not bleed, additional patients who are treated on demand only will be included enabling to study possible modulatory effects of different hemostatic factors (particularly prothrombotic and thrombin activatable fibrinolysis inhibitor (TAFI)) on clinical presentation. The investigators will correlate both those factors and clinical severity with global hemostatic methods.

The investigators expect to prove that individual tailoring of the treatment, which may enable lowering the prophylactic dose of factor concentrate without increasing the risk of bleeding, is justified in some hemophilia patients. This approach would reduce the amount of necessary factor concentrate in certain patients and decrease the cost (which represents extensive burden for health care systems) of treatment without potential risk for the patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with bleeding disorders

Exclusion Criteria:

* none

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients with moderate and severe hA, 30 patients with moderate and severe hB and 50 patients with VWD (primarily severe type I and type III) from hemophilia centers Stockholm, Sweden and Belgrade, Serbia.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2013-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of microparticles | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Antovic JP, Mikovic D, Elezovic I, Holmstrom M, Wilkens M, Elfvinge P, Mahmoud Hourani Soutari N, Antovic A. Two global haemostatic assays as additional tools to monitor treatment in cases of haemophilia A. Thromb Haemost. 2012 Jul;108(1):21-31. doi: 10.1160/TH11-11-0811. Epub 2012 Apr 26. PMID 22534727
- [Result] Mobarrez F, Mikovic D, Antovic A, Antovic JP. Is a decrease of microparticles related to improvement of hemostasis after FVIII injection in hemophilia A patients treated on demand? J Thromb Haemost. 2013 Apr;11(4):697-703. doi: 10.1111/jth.12103. PMID 23231463